CLINICAL TRIAL: NCT03039920
Title: The Effects of Electronic Cigarette Smoking on the Arterial Wall and Endothelial Glycocalyx Properties of Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Assistant Professor, University of Athens
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 698/11-3-15
Record Dates: First submitted 2017-01-28; First posted 2017-02-01 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic cigarette with or without nicotine (Active Comparator): Electronic cigarette assisted cessation program
  Interventions: Other: Electronic cigarette
- Smoker control (Active Comparator): Conventional cigarette smoking continuation
  Interventions: Other: Conventional cigarette

INTERVENTIONS:
Other: Electronic cigarette — Smoking of electronic cigarette
  Arms: Electronic cigarette with or without nicotine
Other: Conventional cigarette — Smoking tobacco cigarette
  Arms: Smoker control

SUMMARY:
Electronic cigarette is proposed as a bridge to smoking cessation. In this study we examine its effects on aortic elasticity, glycocalyx integrity, and exhaled carbon monoxide (CO) concentration and platelet function, both acutely and after 1 month of use.

DETAILED DESCRIPTION:
Two smoker groups matched for age and sex will be assessed:

1. a group of 30 current smokers with no diagnosed cardiovascular disease as the control group for chronic phase
2. a group of 30 current smokers with no diagnosed cardiovascular disease who will be using the electronic cigarette with nicotine for 1 month

In the acute phase all 60 smokers will undergo a "sham" smoking for 7 minutes. Afterwards 30 out of 60 smokers will be randomized to smoke either a normal cigarette or an electronic cigarette with nicotine and after a 60 minute washout period these subjects will be crossed over to the alternate mode of smoking (electronic with nicotine or normal cigarette respectively).

The remaining 30 smokers will be randomized to smoke either a normal cigarette or an electronic cigarette without nicotine and after a 60 minute washout period these subjects will be crossed over to the alternate mode of smoking (electronic without nicotine or normal cigarette respectively.

After the completion of the acute phase all 60 smokers will start the use of an electronic cigarette for one month.

In the acute phase, measurements will be performed at baseline, after sham smoking and after smoking of the normal or electronic cigarette (with or without nicotine). The chronic phase measurements will be performed 1 month after use electronic cigarette with nicotine. Thirty current smokers of similar age and sex will serve as controls and will have measurements at baseline and 1 month after baseline assessment. The nicotine concentration of the electronic cigarette fluid used during both phases will be 12 mg/dL, while the participants will be allowed to use their cigarette of preference in the acute phase. In both phases we will assess a) the aortic pulse wave velocity (PWV) and augmentation index (AIx) by Arteriograph and Complior; b) the perfusion boundary region of the sublingual arterial microvessels using Sideview, Darkfield imaging (Microscan, Glycocheck); c) the exhaled carbon monoxide (CO) level (parts per million -ppm) as a smoking status marker; d) the vital signs; e) an electrocardiogram; and f) plasma levels of C- reactive protein (CRP), transforming growth factor-b (TGF-b), lipoprotein associated phospholipase A2 (LP- LPA2), tumor necrosis factor- α (TNF-α), interleukins 6 and 10 (IL-6 and -10), procollagen propeptide type III (PIIINP), matrix metalloproteinase 2 and 9 (MMP-2 and -9), and macrophage-colony stimulating factor (MCSF), malondialdehyde (MDA) and protein carbonyls (PC) and platelet function tests using the novel Platelet Function Analyzer PFA-100 and the traditional Light Transmission Aggregometry (LTA)

ELIGIBILITY:
Inclusion Criteria:

* Active conventional cigarette smoker

Exclusion Criteria:

* Health condition adversely affected by smoking, history or presence of cardiovascular disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-01-31 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Acute electronic cigarette vaping effects on arterial stiffness. | 7 minutes
  Acute electronic cigarette vaping effects on arterial stiffness as assessed by pulse wave velocity (PWV, m/sec). PWV (m/sec) was measured by using tonometry by Complior (Alam Medical, Vincennes, France). Two non-invasive pressure sensors were used to record the carotid and femoral waveforms and the distance between the two arterial sites was measured with a tape measure.
Acute electronic cigarette vaping effects on endothelial integrity. | 7 minutes
  Acute electronic cigarette vaping effects on endothelial integrity as assessed by measuring endothelial glycocalyx thickness. We measured the perfused boundary region (PBR) of the sublingual arterial microvessels (ranged from 5 to 25 μm) using Sidestream Darkfield Imaging (Microscan, Glycocheck, Microvascular Health Solutions Inc., Salt Lake City, UT, USA).
Chronic electronic cigarette vaping effects on arterial stiffness. | 1 month
  Chronic electronic cigarette vaping effects on arterial stiffness, as assessed by pulse wave velocity (PWV, m/sec). PWV (m/sec) was measured by using tonometry by Complior (Alam Medical, Vincennes, France). Two non-invasive pressure sensors were used to record the carotid and femoral waveforms and the distance between the two arterial sites was measured with a tape measure.
Chronic electronic cigarette vaping effects on endothelial integrity. | 1 month
  Chronic electronic cigarette vaping effects on endothelial integrity as assessed by measuring endothelial glycocalyx thickness. We measured the perfused boundary region (PBR) of the sublingual arterial microvessels (ranged from 5 to 25 μm) using Sidestream Darkfield Imaging (Microscan, Glycocheck, Microvascular Health Solutions Inc., Salt Lake City, UT, USA).
Chronic electronic cigarette vaping effects on platelet aggregation. | 1 month
  Chronic electronic cigarette vaping effects on platelet function as assessed by Light Transmission Aggregometry (LTA). We measured both maximum (peak) and late platelet aggregation (%) (at 6 minutes) after addition of epinephrine (as stimulant) in platelet rich plasma.The 100% line was set using platelet poor plasma and a 0% baseline established with platelet rich plasma before addition of the agonist(epinephrine). Platelet aggregation is experssed as % of the 100% line
Chronic electronic cigarette vaping effects on high-shear stress-dependent platelet function. | 1 month
  Chronic electronic cigarette vaping effects on high-shear stress-dependent platelet function as assesed by PFA-100. The instrument estimates the ability of platelets activated in a high shear environment to occlude an aperture in a membrane coated with collagen and epinephrine (CEPI).The time taken for flow across the membrane to stop (closure time, CT, seconds) is recorded as measure of platelet function. Platelet adhesion and aggregation following a vascular injury is simulated in vitro by PFA.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Dr, Principal Investigator — Attikon Hospital
Locations (1):
- ''Attikon'' University General Hospital, Athens, Attica, Greece

REFERENCES:
- [Derived] Ikonomidis I, Vlastos D, Kourea K, Kostelli G, Varoudi M, Pavlidis G, Efentakis P, Triantafyllidi H, Parissis J, Andreadou I, Iliodromitis E, Lekakis J. Electronic Cigarette Smoking Increases Arterial Stiffness and Oxidative Stress to a Lesser Extent Than a Single Conventional Cigarette: An Acute and Chronic Study. Circulation. 2018 Jan 16;137(3):303-306. doi: 10.1161/CIRCULATIONAHA.117.029153. No abstract available. PMID 29335291